CLINICAL TRIAL: NCT06428175
Title: Hospital-to-Home Care Coordination for Children and Youth With Special Health Care Needs
Brief Title: Hospital-to-Home Transitional Care Interventions (H2H-TCI) Children/Youth With Special Health Care Needs (CYSHCN)
Acronym: H2H-CYSHCN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00114934
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Health Care; Pediatrics; Transitional Care; Comparative Effectiveness; Family Engagement
Keywords: Special Needs; Hospital to Home Care; Children and Youth with Special Health Care Needs; Randomized Trial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused Dose Hospital-to-Home Transitional Care Interventions (Active Comparator)
  Interventions: Behavioral: Focused Dose Hospital-to-Home Transitional Care Interventions
- Extended Dose Hospital-to-Home Transitional Care Interventions (Active Comparator)
  Interventions: Behavioral: Extended Dose Hospital-to-Home Transitional Care Interventions

INTERVENTIONS:
Behavioral: Focused Dose Hospital-to-Home Transitional Care Interventions — Focused dose H2H-TCIs will consist of a one-time post-discharge phone call completed within 72 hours post-hospital discharge by a clinical interventionist (e.g., nurse care coordinator or care manager). Calls will follow a structured template that provides empirically supported core H2H-TCI functions (follow-up care access, contingency planning, medication review, family education). The interventionist will also conduct a pre-hospital discharge clinical needs assessment with the parent.
  Arms: Focused Dose Hospital-to-Home Transitional Care Interventions
Behavioral: Extended Dose Hospital-to-Home Transitional Care Interventions — Extended dose H2H-TCIs will include a pre-discharge clinical needs assessment and initial phone call within 72 hours post-discharge, similar to the focused arm. After the initial contact, the dose of the extended H2H-TCI will increase as subjects receive high-intensity support during weekly post-discharge phone contacts through 30 days post-discharge. All contacts in the extended dose arm will be completed by a transition coach interventionist (e.g., nurse care coordinator or care manager) who will be formally trained on pillars of the Care Transitions Intervention© (CTI), a multi-faceted H2H-TCI that is the basis for the extended dose arm.
  Arms: Extended Dose Hospital-to-Home Transitional Care Interventions

SUMMARY:
Aim 1: Compare the effectiveness of focused dose vs extended dose hospital-to-home Transitional Care Interventions (H2H-TCI) on health service use and parent-reported confidence for hospitalized CYSHCN. Aim 2: Compare the effectiveness of focused and extended dose H2H-TCI among vulnerable CYSHCN subgroups. Hypothesis: Both H2H-TCI arms will improve primary outcomes more for CYSHCN with higher versus lower clinical complexity; while extended H2H-TCI will better mitigate racial/ethnic outcome disparities than focused H2H-TCI. Aim 3: Evaluate implementation context, processes, and mechanisms via a multi-phase mixed methods study design.

DETAILED DESCRIPTION:
Primary Aims Aim 1: Compare the effectiveness of focused dose vs extended dose hospital-to-home Transitional Care Interventions (H2H-TCI) on health service use and parent-reported confidence for hospitalized CYSHCN.

Hypothesis: Extended H2H-TCI will be associated with lower acute care use and higher confidence than focused H2H-TCI.

Secondary Aims Aim 2: Compare the effectiveness of focused and extended dose H2H-TCI among vulnerable CYSHCN subgroups.

Hypothesis: Both H2H-TCI arms will improve primary outcomes more for CYSHCN with higher versus lower clinical complexity; while extended H2H-TCI will better mitigate racial/ethnic outcome disparities than focused H2H-TCI.

Aim 3: Evaluate implementation context, processes, and mechanisms via a multi-phase mixed methods study design.

The study populations consist of adult parent/caregivers' dyad and children/youth with special health care needs. Participants will be randomized to focused dose intervention after discharge or an extended dose intervention. the single dose will receive one phone call from an interventionist post discharge, the extended dose group will receive weekly phone calls for one month from an interventionist.

Analysis of data from the confidence-mediated and vulnerable patient/family characteristics-moderated pathways will address Aims 1 and 2, respectively.

During extraction of data from each site's Electronic Health Record (EHR) data security risks will be mitigated by following established standard operating procedures at Duke and the University of North Carolina (UNC). During preparation of site-based analytical datasets risks will be mitigated by limiting Protected Health Information (PHI) as much as and as early as is practical. All datasets will be stored and reviewed on a secure, cloud-based Protected Analytical and Computing Environment (PACE) at Duke and at UNC in the Secure Research Workspace (SRW).

The investigators will plan to create a Data Safety and Monitoring Board (DSMB) that includes expert clinicians who are not active study team members and are independent of the study sponsor. The DSMB will oversee the safety of volunteers participating in the study as needed.

ELIGIBILITY:
Inclusion Criteria:

* For this study, eligible children/youth with special health care needs (CYSHCN) and adult parent/caregiver dyads will be those who meet the following inclusion criteria:

  1. Child is a CYSHCN, defined as having seen two or more distinct specialty areas for outpatient visits during the 12 months prior to index hospitalization admission date
  2. Age of hospitalized child is under 18 years old
  3. Child hospitalized on a general pediatrics inpatient service line at participating site
  4. Adult parent/caregiver for the child is 18 years or older

Exclusion Criteria:

* Child exclusion criteria:

  1. Child will be discharged to any location besides home (e.g., long-term care or residential facility, skilled nursing facility, inpatient acute rehabilitation, psychiatric facility)
  2. Child is a ward of the state or has an ongoing social services investigation
  3. Child is already receiving transitional care, intensive longitudinal care coordination (e.g., organ/disease-specific clinical program, clinical division within the same institution as the hospital [e.g., Children's Complex Care Program at UNC; Complex Care Service at Duke]), and/or longitudinal population health care coordination as part of a bundled alternative payment care model.
* Parent/caregiver exclusion criteria include:

  1. Age less than 18 years old
  2. Diminished capacity to provide consent/participate
  3. Primary language for parent/caregiver is any language besides English or Spanish

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
30-day acute care use | 30 days post-hospital discharge
  30-day, all-cause composite readmission and emergency department (ED) visit rate
Caregiver confidence | Baseline, 30 days post-discharge
  Change in caregiver-reported confidence that their child can avoid hospitalization within the next one month (1=not confident; 10=fully confident; <5 is low confidence)

SECONDARY OUTCOMES:
7-day acute care use | 7-days post-discharge
  All-cause composite readmission and ED visit rate at 7 days
14-day acute care use | 14 days post-discharge
  All-cause composite readmission and ED visit rate at 14 days
Readmissions | 7, 14, 30 days post-discharge
  All-cause readmission rate at 7, 14, and 30 days
Emergency Department (ED) visits | 7, 14, 30 days post-discharge
  All-cause ED visits at 7, 14, and 30 days
Outpatient follow-up visit attendance | 7, 14, 30 days post-discharge
  Completed outpatient visits by clinical area (primary, specialty, allied health)
Days at home | 30 and 90 days post-discharge
  Annualized days without clinical visits (clinical days without healthcare visits)
Caregiver strain | Baseline, 7, 14, 30, and 90-days post-discharge
  Change in caregiver-reported strain (measured by scores on seven-item Caregiver Strain Questionnaire Short Form 7, CGSQ-SF7 survey), where a higher score indicates a higher level of caregiver strain.
Global health status | Baseline, 7, 14, 30, and 90-days post-discharge
  Change in caregiver-reporter PROMIS global health status survey. PROMIS assessments are scored on a T-score metric. High scores mean more of the concept being measured. 10 points on the T-score metric is one standard deviation (SD). PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population.
Caregiver mental health-related quality of life (HR-QOL) | Baseline, 7, 14, 30, and 90-days post-discharge
  Change in caregiver-reported mental HR-QOL as scored on the Medical Outcomes Short Form 12 (SF12) survey.
Quality of hospital-to-home care transitions | 30 days post-discharge
  Pediatric Transition Experience Measure (P-TEM): eight-item, parent-reported measure of overall process and quality of hospital-to-home transitions.
Fidelity | approximately 90 days post-discharge
  Percentage of intervention core components delivered as planned (goal: ≥80%)
Feasibility Acceptability Appropriateness | approximately 90 days post-discharge
  Clinical staff and caregiver-reported composite score responses to Feasibility of Implementation, Acceptability of Implementation, and Implementation Appropriateness surveys (4 items each)

CONTACTS AND LOCATIONS:
Overall Officials: David Ming, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - UNC Hospitals, Chapel Hill, North Carolina
  - DUHS, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No